CLINICAL TRIAL: NCT05140850
Title: Long-term Consequences of Neuroimaging and Perceived Cognitive Dysfunction in Obstetrics Posterior Reversible Encephalopathy Syndrome
Brief Title: Long-term Consequences of Neuroimaging and Perceived Cognitive Dysfunction in oPRES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Director of obstetrics, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: 82001568
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Neuroimaging; Cognitive Dysfunction; Posterior Reversible Encephalopathy Syndrome
MeSH Terms: conditions — Cognitive Dysfunction; Posterior Leukoencephalopathy Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRES group: PE or E with PRES
  Interventions: Biological: neuroimaging examination,neuro-cognitive test,blood pressure,blood sample
- non-PRES group: PE or E without PRES
  Interventions: Biological: neuroimaging examination,neuro-cognitive test,blood pressure,blood sample

INTERVENTIONS:
Biological: neuroimaging examination,neuro-cognitive test,blood pressure,blood sample — neuroimaging will be perform,neuro-cognitive will be tested,blood pressure will be monitored,blood samples will be tested

SUMMARY:
The purpose of this study is to explore the long-term consequences of neuroimaging and perceived cognitive dysfunction in obstetrics posterior reversible encephalopathy syndrome.

DETAILED DESCRIPTION:
This is a prospective study. The investigators divided the PE or E patients into two groups, namely PRES group and non-PRES group, according to diagnostic criteria . The general information（demographic data，blood pressure.etc.）and blood sample will be collected. Additionally,all patients receive neuroimaging examination（DTI,ASL,3D-TMI.etc.）and neuro-cognitive test（MMSE,MOCA,CFQ, etc.） to assess the cerebral white matter lesions and cognitive changes.

ELIGIBILITY:
Inclusion Criteria:

1. patients were diagnosed of PE or E
2. patients received cranial image examination
3. patients consent to participate

Exclusion Criteria:

1. patients combined other neurological diseases
2. patients combined mental illness

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We divided the PE or E patients into two groups, namely PRES group and non-PRES group, according to diagnostic criteria . the general information（demographic data，blood pressure.etc.）and blood sample will be collected.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
neuroimaging examination | within 10 years after deliver
  the degree of white matter lesions(0,normal; 1, limited cortical or subcortical white matter oedema; 2, white matter oedema > cortical oedema, white matter oedema extending into deep white matter; 3, white matter oedema > cortex oedema, oedema extending to the ventricular surface; 4, the involved regions substantially extend to the ventricular surface and are almost completely conﬂuent; 5, involved regions are fully conﬂuent and continuous, ventricular deformity due to the oedema).The value of fractional anisotropy(FA) in PRES group may higher than non- PRES group, and mean diffusivity (MD) in PRES group may lower than non- PRES group.
neuro-cognitive test of Mini-mental State Examination | within 10 years after deliver
  the scores of Mini-mental State Examination,normal (27-30);mild (21-26); moderate (10-20); severe (0-9).
neuro-cognitive test of Montreal Cognitive Assessment | within 10 years after deliver
  the scores of Montreal Cognitive Assessment,normal (≥26); abnormal (<26).
blood pressure and hypertension | within 10 years after deliver
  Hypertension: blood pressure ≥140/90 mmHg
level of lactate dehydrogenase(LDH) | within 10 years after deliver
  inflammatory: LDH>380U/L
level of LDL in blood | within 10 years after deliver
  hyperlipidemia：LDL>3.12mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No